CLINICAL TRIAL: NCT03682653
Title: Neonates and Azithromycin, an Innovation in the Treatment of Children in Burkina Faso
Acronym: NAITRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OPP1187628-B
Record Dates: First submitted 2018-09-19; First posted 2018-09-24 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Childhood Mortality
Keywords: childhood mortality; neonates; azithromycin; mass drug administration
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: individually randomized trial of azithromycin versus placebo to establish the efficacy and safety of administration of a dose of azithromycin during the neonatal period
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithromycin (Active Comparator): a single dose of Azithromycin will be administered to infants between their 8-27th days of life
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): a single dose of placebo will be administered to infants between their 8-27th days of life
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — a single dose of Azithromycin will be administered to infants between their 8-27th days of life
  Arms: Azithromycin
Drug: Placebo — a single dose of Placebo will be administered to infants between their 8-27th days of life
  Arms: Placebo

SUMMARY:
Although under-5 mortality rates are declining globally, neonatal mortality remains persistently high in many regions of sub-Saharan Africa. Mass azithromycin distribution to children aged 1-59 months has been shown to reduce childhood mortality in Niger, Tanzania, and Malawi. This study did not evaluate the effect of azithromycin administered during the neonatal period. Observational evidence from high income countries has suggested that macrolides, including erythromycin and azithromycin, may be associated with increased risk of development of infantile hypertrophic pyloric stenosis (IHPS). However, these studies are limited by confounding by indication, as infants only receive antibiotics when they are ill.

The investigators proposed an individually randomized trial of azithromycin versus placebo to establish the efficacy and safety of administration of a dose of azithromycin during the neonatal period. The long-term goal is generate evidence that can be used by neonatal and child survival programs related to the use of azithromycin in the youngest children who have the highest risk of mortality. The investigators hypothesize that a single dose of azithromycin administered in the neonatal period will lead to significantly reduced risk of mortality and that this dose will be safe.

Objectives

1. Establish the efficacy of a single dose of azithromycin administered during the neonatal period compared to placebo in infants 8 to 27 days of life for reduction in all-cause mortality.
2. Establish the safety of a single dose of azithromycin administered during the neonatal period.

This study will be conducted in several regions of Burkina Faso, including peri-urban areas of Ouagadougou and Nouna town, and rural areas that are within 4 hours' drive of a pediatric facility with capacity for performing pyloromyotomy

DETAILED DESCRIPTION:
Child mortality in West Africa is among the highest in the world. Although child health and mortality are improving worldwide, children in the Sahel and sub-Sahel regions of West Africa have the greatest risks of mortality. Burkina Faso's current under-5 mortality rate is estimated 110 per 1,000 live births. Similar to other countries in the region, the major causes of child mortality in Burkina Faso are malaria, respiratory tract infection, and diarrhea. Malnutrition acts as a major underlying contributor to mortality. Neonatal mortality remains persistently high, with approximately 1/5th of neonatal mortality due to pneumonia, meningitis, and sepsis. Interventions that address these underlying causes may be particularly efficacious for reducing mortality.

Younger children at are at a higher risk of mortality. Approximately 2/3rd of under-5 deaths occur during the first year of life. In general, the child mortality rate decreases as age increases. While some improvement has been observed, neonatal mortality is declining at a slower rate than post-neonatal childhood mortality. Many child health interventions are designed specifically for children over 6 months of age, such as vitamin A supplementation, seasonal malaria chemoprevention, and lipid-based nutritional supplementation. Identification of strategies that are safe and effective for the youngest children will be required to address persistently high rates of neonatal and infant mortality.

The MORDOR I study demonstrated a significant reduction in all-cause child mortality following biannual mass azithromycin distribution. Across three diverse geographic locations in sub-Saharan Africa (Malawi, Niger, and Tanzania), biannual mass azithromycin distribution over a two-year period led to a 14% decrease in all-cause child mortality. In Niger, 1 in 5-6 deaths were averted. These results are qualitatively similar to those of a previous study of mass azithromycin distribution for trachoma control in Ethiopia, which found reduced odds of all-cause mortality in children in communities receiving mass azithromycin compared to control communities.

In MORDOR I, the strongest effect of azithromycin was in the youngest cohort of children. Across all three countries, the strongest effect of azithromycin was consistently in children 1-5 months of age, with an approximately 25% reduction in all-cause mortality. However, MORDOR I was not optimized to target the youngest age groups. Although children as young as 1 month were eligible, biannual distributions might not reach some children until 7 months of age. On average, children were first treated at 4 months. Given that there may be a substantial benefit to treating children at younger ages, azithromycin strategies that are designed to target younger age groups may be even more beneficial for reducing child mortality.

Here, the investigators propose a randomized controlled trial designed to evaluate the efficacy of a dose of azithromycin administered during the neonatal period for prevention of mortality within in the first 6 months of life. The investigators propose to randomize births in several geographic regions of Burkina Faso to a single dose of azithromycin or placebo between day 8 and 27 of life. This study is designed to provide evidence of the efficacy of azithromycin treatment for the youngest children.

ELIGIBILITY:
Communities

Inclusion Criteria:

* Within 4 hours of a facility that can provide services for pyloromyotomy (Ouagadougou or Bobo Dioulasso)
* Accessible during the rainy season
* Ultrasound machine available OR a facility in which an ultrasound machine could be placed is within 1 hour

Exclusion Criteria:

* Refusal of village chief

Individuals:

Inclusion Criteria:

* Weight over 2500 g
* Able to feed orally
* Family intends to stay in study area for at least 6 months
* Appropriate consent from at least one caregiver
* No known allergy to azalides
* Not living within one of the communities included in the community study(CHAT/CHATON)
* No hepatic failure manifested by neonatal jaundice

Exclusion Criteria:

* Weight <2500 g
* Unable to feed orally
* Family planning to move
* Mother/caregiver not willing to participate
* Allergic to azalides
* Living in one of the communities included in the community study (CHAT/CHATON)
* Hepatic failure manifested by neonatal jaundice

Ages: 8 Days to 27 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21832 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Oldenburg, PhD, Principal Investigator — University of California, San Francisco; Tom M Lietman, MD, Principal Investigator — University of California, San Francisco; Ali Sie, MD, PhD, Principal Investigator — Centre de Recherche en Sante de Nouna, Burkina Faso
Locations (1):
- Centre de Recherche En Santé de Nouna, Nouna, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available as per the Bill and Melinda Gates open access policy. Individual participant data will be available that underline the reported results (texts, tables, figures, and appendices). The study protocol and statistical analysis plan will also be made available. The data will be available following publication in accordance with the BMGF guidelines.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available following publication, without any embargo period.

REFERENCES:
- [Derived] Bountogo M, Sie A, Zakane A, Compaore G, Ouedraogo T, Brogdon J, Lebas E, Nyatigo F, Medvedev MM, Arnold BF, Lietman TM, Oldenburg CE; NAITRE Study Team. Infant mortality and growth failure after oral azithromycin among low birthweight and underweight neonates: A subgroup analysis of a randomized controlled trial. PLOS Glob Public Health. 2023 May 15;3(5):e0001009. doi: 10.1371/journal.pgph.0001009. eCollection 2023. PMID 37186577
- [Derived] Sie A, Bountogo M, Zakane A, Compaore G, Ouedraogo T, Ouattara M, Lebas E, Brogdon J, Nyatigo F, O'Brien KS, Porco TC, Barnighausen T, Arnold BF, Lietman TM, Oldenburg CE; NAITRE Study Team. Neonatal Azithromycin Administration and Growth during Infancy: A Randomized Controlled Trial. Am J Trop Med Hyg. 2023 Mar 27;108(5):1063-1070. doi: 10.4269/ajtmh.22-0763. Print 2023 May 3. PMID 36972694
- [Derived] Oldenburg CE, Sie A, Bountogo M, Zakane A, Compaore G, Ouedraogo T, Koueta F, Lebas E, Brogdon J, Nyatigo F, Doan T, Porco TC, Arnold BF, Lietman TM; NAITRE Study Team. Neonatal azithromycin administration for prevention of infant mortality. NEJM Evid. 2022 Apr;1(4):EVIDoa2100054. doi: 10.1056/EVIDoa2100054. Epub 2022 Mar 17. PMID 35692260
- [Derived] Bountogo M, Sie A, Zakane A, Compaore G, Ouedraogo T, Lebas E, Brogdon J, Nyatigo F, Arnold BF, Lietman TM, Oldenburg CE. Antenatal care attendance and risk of low birthweight in Burkina Faso: a cross-sectional study. BMC Pregnancy Childbirth. 2021 Dec 13;21(1):825. doi: 10.1186/s12884-021-04310-6. PMID 34903190
- [Derived] Sie A, Bountogo M, Nebie E, Ouattara M, Coulibaly B, Bagagnan C, Zabre P, Lebas E, Brogdon J, Godwin WW, Lin Y, Porco T, Doan T, Lietman TM, Oldenburg CE; NAITRE Study Group. Neonatal azithromycin administration to prevent infant mortality: study protocol for a randomised controlled trial. BMJ Open. 2019 Sep 4;9(9):e031162. doi: 10.1136/bmjopen-2019-031162. PMID 31488494

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azithromycin | Placebo
Started | 10898 | 10934
Received Allocated Treatment | 10898 | 10928
Day 21 | 10069 | 10119
3 Months | 10273 | 10356
Completed (6 Months (primary endpoint)) | 9606 | 9684
Not Completed | 1292 | 1250

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Total
Number analyzed (Participants) | 10898 | 10934 | 21832
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 11 [9 to 15] | 11 [9 to 14] | 11 [9 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5413 | 5431 | 10844
  Male | 5485 | 5503 | 10988
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Burkina Faso: Center | 919 | 951 | 1870
  Burkina Faso: Boucle du Mouhoun | 1299 | 1329 | 2628
  Burkina Faso: Cascade | 2009 | 1977 | 3986
  Burkina Faso: Center Ouest | 1217 | 1211 | 2428
  Burkina Faso: Hauts-Bassins | 5454 | 5465 | 10919
  Burkina Faso: Missing | 0 | 1 | 1
Urban dwelling [Count of Participants; unit: Participants]
  Urban | 8960 | 9055 | 18015
  Rural | 1932 | 1869 | 3801
  Missing | 6 | 10 | 16
Season of enrollment [Count of Participants; unit: Participants]
  Rainy (June to October) | 5217 | 5295 | 10512
  Dry (November to May) | 5681 | 5639 | 11320
Birthweight [Median (Inter-Quartile Range); unit: g] | 3000 [2700 to 3250] | 3000 [2700 to 3260] | 3000 [2700 to 3250]
Weight at enrollment [Median (Inter-Quartile Range); unit: g] | 3300 [2980 to 3620] | 3300 [2990 to 3620] | 3300 [2990 to 3620]
Length at enrollment [Median (Inter-Quartile Range); unit: cm] | 50.4 [49.3 to 51.9] | 50.5 [49.3 to 52.0] | 50.5 [49.3 to 51.9]
Wasted [Count of Participants; unit: Participants] — Defined as Weight-for-length Z-score (WLZ) < -2 SD.
  Participants | 531 | 559 | 1090
Underweight [Count of Participants; unit: Participants] — Defined as Weight-for-age Z-score (WAZ) < -2 SD.
  Participants | 658 | 652 | 1310
Stunted [Count of Participants; unit: Participants] — Defined as Length-for-age Z-score (LAZ) < -2 SD.
  Participants | 884 | 869 | 1753
MUAC [Median (Inter-Quartile Range); unit: cm] — mid-upper-arm circumference; MUAC < 12.5 cm indicates Moderate acute malnutrition
  cm | 10.9 [10.0 to 11.5] | 11.0 [10.0 to 11.5] | 11.0 [10.0 to 11.5]
Mother's age [Median (Inter-Quartile Range); unit: years] | 25 [21 to 30] | 25 [21 to 30] | 25 [21 to 30]
Mother's education [Count of Participants; unit: Participants]
  None | 5910 | 6029 | 11939
  Primary | 1990 | 1978 | 3968
  Secondary or above | 2997 | 2923 | 5920
  Missing | 1 | 4 | 5
No. children in household [Median (Inter-Quartile Range); unit: children] | 1 [0 to 3] | 1 [0 to 3] | 1 [0 to 3]
Pregnancy type [Count of Participants; unit: Participants]
  Singleton | 10702 | 10753 | 21455
  Multiple | 195 | 177 | 372
  Missing | 1 | 4 | 5
No. of antenatal visits [Median (Inter-Quartile Range); unit: visits] | 4 [3 to 5] | 4 [3 to 5] | 4 [3 to 5]
Initiation of breastfeeding [Count of Participants; unit: Participants]
  Immediate | 10320 | 10341 | 20661
  Delayed | 566 | 574 | 1140
  Not breastfeeding | 11 | 15 | 26
  Missing | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Mortality - All Cause
Description: The primary outcome of the study was all-cause mortality rate in infants at 6 months of age.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 9606 | 9684
Participants | 42 | 50

2. Secondary Outcome: 12 Month Mortality - All Cause
Description: All-cause Mortality Rate in infants at 12 months of age
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 9534 | 9563
Participants | 52 | 64

3. Secondary Outcome: Vital Status
Description: Caregivers will be asked if the child is dead or alive at 365 days of life
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 9534 | 9563
Participants | 52 | 64

4. Secondary Outcome: Change in Weight Over Time
Description: Weight gain from baseline to day 180
Time Frame: 6 months
Population: 1 missing weight measure at baseline in placebo arm.
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 9475 | 9626
g/day | 23.2 (5.3) | 23.3 (5.4)

5. Secondary Outcome: Change in Length Over Time
Description: Change in length from baseline to day 180
Time Frame: 6 months
Population: 4 missing length measures at baseline. All in placebo arm.
Measure: Mean (Standard Deviation); unit: mm/day
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 9475 | 9623
mm/day | 0.9 (0.2) | 0.9 (0.2)

6. Secondary Outcome: Proportion of Infants Developing Infantile Hypertrophic Pyloric Stenosis
Description: Proportion of infants developing infantile hypertrophic pyloric stenosis between 2 to 8 weeks after treatment
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 10898 | 10934
Participants | 1 | 0

7. Secondary Outcome: Adverse Events
Description: Caregivers will be asked if their child experienced any symptoms for pyloric stenosis since the last visit.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 9634 | 9643
Participants | 0 | 0

8. Secondary Outcome: Neonatal Mortality
Description: Mortality prior to 28 days of life
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 10485 | 10547
Participants | 9 | 6

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Azithromycin | Placebo
All-Cause Mortality (participants affected / at risk) | 52/10898 | 64/10934
Serious Adverse Events (participants affected / at risk) | 29/10898 | 15/10934
Other Adverse Events (participants affected / at risk) | 575/10898 | 599/10934
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=10898) | Placebo (N=10934)
Infantile hypertrophic pyloric stenosis (Gastrointestinal disorders) | 1 | 0
Hospitalization within 28 d of treatment (General disorders) | 14 | 7
Mortality within 28 d of treatment (General disorders) | 16 | 8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=10898) | Placebo (N=10934)
Vomiting (any) (Gastrointestinal disorders) | 78 | 49
Vomiting after every feed (Gastrointestinal disorders) | 22 | 9
Projectile vomiting (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 51 | 61
Fever (General disorders) | 193 | 237
Abdominal pain (General disorders) | 209 | 171
Rash (Skin and subcutaneous tissue disorders) | 70 | 86
Constipation (Gastrointestinal disorders) | 82 | 111

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT03682653/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT03682653/SAP_001.pdf